CLINICAL TRIAL: NCT03248466
Title: Transplantation of Autologous Platelet Rich Gel Combined With Autologous Bone Marrow Mesenchymal Stem Cells for Treatment of Diabetic Foot Ulcer
Brief Title: PRG Combined With Autologous BMMSCs for Treatment of Diabetic Foot Ulcer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Wu Qinan, Doctor, Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: endocrine department of TMMU
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Diabetic Foot Ulcer
Keywords: platelet rich gel; BMMSCs; diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: diabetic foot ulcer which Wagner classification at 2-3 grade.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional treatment (Placebo Comparator): Traditional treatment such as insulin,antidiabetes,dressing
  Interventions: Biological: PRG combined with BMMSCs transplantation
- PRG combined with BMMSCs transplantation (Experimental): Traditional treatment such as insulin,antidiabetes,dressing and Autologous PRG combined with BMMSCs
  Interventions: Biological: PRG combined with BMMSCs transplantation
- PRG treatment (No Intervention): Traditional treatment such as insulin,antidiabetes,dressing and Autologous PRG

INTERVENTIONS:
Biological: PRG combined with BMMSCs transplantation — PRG combined with BMMSCs transplantation
  Other Names: PRG
  Arms: PRG combined with BMMSCs transplantation; Traditional treatment

SUMMARY:
To investigate the treatment effect between Traditional treatment and transplantation of autologous PRG combined with autologous BMMSCs for treatment of diabetic foot ulcer.

DETAILED DESCRIPTION:
60 diabetic foot ulcer in our hospital will divide into 3 groups: group A (20 diabetic foot ulcer who give Traditional treatment), group B (20 diabetic foot ulcer who give Traditional treatment and transplantation of autologous platelet rich gel)，group C (20 diabetic foot ulcer who give Traditional treatment and transplantation of autologous platelet rich gel combined with autologous bone marrow mesenchymal stem cells). The age, height, weight, blood glucose, glycosylated hemoglobin A1c（HbA1c）, lipid, blood pressure, course of disease, Wound healing rate,transcutaneous oxygen pressure,Amputation rate,Hospital stay will record respectively. And High-sensitive C-reactive protein (HsCRP) and Tumor necrosis factor-α（TNF-α） will detect as Baseline. After each group's treatment, Change from baseline of all indexes will record, one way Analysis of Variance will be analyzed the significantion among 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic foot according to The Wagner is 2-3 graded;

Exclusion Criteria:

* Type 1 diabetes mellitus,presence of autoimmune diabetes;
* Gestational diabetes;
* Patients with heart, liver, or renal function impairment;presence of severe infections or cerebrovascular disease.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-30 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Amputation rate | up to 6 months
  Amputation rate up to 6 months
hospital stay | up to 6 months
  hospital stay

SECONDARY OUTCOMES:
Wound healing time | up to 6 months
  Wound healing time
Transcutaneous oxygen partial pressure | Transcutaneous oxygen partial pressure up to 6 months
  Transcutaneous oxygen partial pressure

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Southwest Hospital of the Third Military Medical University, Chongqing, Chongqing Municipality
  - Endocrine Department, the First Affiliated Hospital of the Third Military Medical University, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No